CLINICAL TRIAL: NCT01206257
Title: This is an International, Prospective, Non-interventional Study, Company Sponsored, Multi-center Study. Patients Undergo Coronary Angiography or PCI Procedure With Ultravist. The Primary Objective is to Evaluate the Safety and Tolerability.
Brief Title: The Safety and toleRability of UltraviSt in Patients Undergoing Cardiac CaTheterization (TRUST)
Acronym: TRUST
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Director, Bayer Healthcare AG
Other Study IDs: 15454; UV1010CN (Other: company internal)
Record Dates: First submitted 2010-09-20; First posted 2010-09-21 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Angiocardiography
Keywords: Survey; Angiography; ADR; Image quality
MeSH Terms: interventions — iopromide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Iopromide (Ultravist, BAY86-4877)

INTERVENTIONS:
Drug: Iopromide (Ultravist, BAY86-4877) — Intravenous/intraarterial digital subtraction angiography (DSA); Generally doses of up to 1.5 g iodine per kg body weight are well tolerated.

SUMMARY:
This study is to collect the information of Ultravist® in the patients indicated for the coronary angiography or PCI, like rate of ADR in patients, the dose for different indications, image quality to prove Ultravist the good safety and effectivity

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients who receive Ultravist® for coronary angiography or PCI can be included in the study

Exclusion Criteria:

* Patients who are or are suspected in pregnancy or nursery
* Patients with the contraindications for Ultravist
* Patients with the contraindications for cardiac catheterization

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who plan to undergo coronary angiography or PCI procedure with ultravist will be enrolled
Sampling Method: Probability Sample
Enrollment: 17513 (Actual)
Dates: Start 2010-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of the safety and tolerability of Ultravist® in patients Undergoing cardiac catheterization. | 12 months

SECONDARY OUTCOMES:
Estimation of the image quality of Ultravist® | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, China